CLINICAL TRIAL: NCT05370313
Title: ETM Taxes Study 1: The Impact of Innovative Tax Proposals on Purchase Patterns
Brief Title: The Impact of Innovative Tax Proposals on Purchase Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Roswell Park Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Stein, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VT IRB # 22-433
Record Dates: First submitted 2022-04-29; First posted 2022-05-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — metariboadenosine triphosphorous

STUDY DESIGN:
Intervention Model Description: Participants will each complete two control trials and four Experimental Marketplace conditions, representing each of the four tax proposals. The order of tax proposal conditions will be determined randomly. Within each condition, taxes will be increased proportionally across 5 trials to examine how cigarette purchasing, substitution, and poly-tobacco purchasing (i.e., diversity in products purchased) are affected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cigarette smokers - Sequence 1 (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and each of the four tax policy conditions in this sequence: Tobacco Parity, Modified Risk Tobacco Products, Harm Reduction, Nicotine Content.
  Interventions: Behavioral: Market Price Condition (control); Behavioral: Tobacco Parity Tax Condition; Behavioral: Nicotine-Content Tax Condition; Behavioral: Harm-Reduction Tax Condition; Behavioral: Modified Risk Tobacco Product (MRTP) Tax Condition
- Cigarette smokers - Sequence 2 (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and the four tax policy conditions in this sequence: Nicotine Content, Tobacco Parity, Modified Risk Tobacco Products, Harm Reduction.
  Interventions: Behavioral: Market Price Condition (control); Behavioral: Tobacco Parity Tax Condition; Behavioral: Nicotine-Content Tax Condition; Behavioral: Harm-Reduction Tax Condition; Behavioral: Modified Risk Tobacco Product (MRTP) Tax Condition
- Cigarette smokers - Sequence 3 (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and each of the the four tax policy conditions in this sequence: Modified Risk Tobacco Products, Harm Reduction, Nicotine Content, Tobacco Parity.
  Interventions: Behavioral: Market Price Condition (control); Behavioral: Tobacco Parity Tax Condition; Behavioral: Nicotine-Content Tax Condition; Behavioral: Harm-Reduction Tax Condition; Behavioral: Modified Risk Tobacco Product (MRTP) Tax Condition
- Cigarette smokers - Sequence 4 (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to two control trials and each of the the four tax policy conditions in this sequence: Harm Reduction, Nicotine Content, Tobacco Parity, Modified Risk Tobacco Products.
  Interventions: Behavioral: Market Price Condition (control); Behavioral: Tobacco Parity Tax Condition; Behavioral: Nicotine-Content Tax Condition; Behavioral: Harm-Reduction Tax Condition; Behavioral: Modified Risk Tobacco Product (MRTP) Tax Condition

INTERVENTIONS:
Behavioral: Market Price Condition (control) — Nicotine/tobacco products available in the Experimental Tobacco Marketplace at market price. Cigarette taxes increased across trials at the same magnitudes used in the tax conditions.
Behavioral: Tobacco Parity Tax Condition — Tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all tobacco products are placed in the high-tax tier while products that do not contain tobacco (e.g., herbal cigarettes and nicotine-free ENDS) are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier.
Behavioral: Nicotine-Content Tax Condition — Tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, products with greater than 3 mg nicotine per single unit are placed in the high-tax tier, products with 0.6-3.0 mg/unit in the medium-tax tier, and those with 0.5 mg/unit or less in the no-tax tier.
Behavioral: Harm-Reduction Tax Condition — Tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all combustible products with high abuse liability are placed in the high-tax tier. All non-combustible products or combustible products with low abuse liability are placed in the medium-tax tier. Nicotine Replacement Therapy products are placed in the no-tax tier.
Behavioral: Modified Risk Tobacco Product (MRTP) Tax Condition — Tobacco products in the Experimental Tobacco Marketplace are placed into three tax tiers: high-, medium-, and no-tax. In this condition, all non-MRTP tobacco products are placed in the high-tax tier, MRTPs are placed in the medium-tax tier, and Nicotine Replacement Therapy products are placed in the no-tax tier.

SUMMARY:
This study will investigate the effect of four tax proposals (i.e. Tobacco Parity, Nicotine-Content, Harm-Reduction, and Modified Risk Tobacco Product-related taxes) on tobacco product purchasing patterns.

DETAILED DESCRIPTION:
This study experimentally examines the effects of largely untried integrated tax proposals. Four tax proposals will be modeled: Tobacco Parity, Nicotine-Content, Harm-Reduction, and MRTP. Tobacco products are placed into three tax tiers: high-, medium-, and no-tax, according to the goals of each proposal. In a within-subjects design, cigarette smokers will complete two control (market price) trials and four conditions in the Experimental Tobacco Marketplace, representing each of the four tax proposals. Within each condition, taxes will be increased proportionally across 5 trials (relative to tax tier) to examine how cigarette purchasing, substitution, and poly-tobacco purchasing (i.e., diversity in products purchased) are affected.

ELIGIBILITY:
Inclusion Criteria:

* provide informed consent
* provide a breath carbon monoxide sample ≥ 8 ppm,
* be at least 21 years of age (the legal age to purchase tobacco),
* smoke at least 10 cigarettes daily, and
* use other tobacco products less than weekly.

Exclusion Criteria:

* report uncontrolled physical or mental health conditions (e.g., uncontrolled diabetes, high blood pressure, major depressive disorder, etc.),
* use of smoking cessation medications (e.g., nicotine replacement, bupropion, varenicline) in the past 30 days,
* report concrete, immediate plans to alter/quit using their usual tobacco products in the next 30 days,
* be pregnant or lactating, or
* have plans to move out of the area during the experiment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Quantity of Tobacco Products Purchased in the High-Tax Tier - Product demand (intensity and elasticity) | 1 day
  Purchasing of high-tax tier products in the ETM conditions will be fit to a commonly used exponential demand model that quantifies the relationship between the multiplicative tax factor (e.g., 2 times base tax rate) and purchasing of high-tax tier products. This demand analysis (which assumes a negative association between price and purchasing) will be used in the high-tax tier products because participants will be conventional cigarette smokers and these products (when available) will always be in that tier. As such, we expect participants to defend their purchase of cigarettes in the high-tax tier under a variety of conditions. Demand estimates will be obtained for each participant in each tax proposal.
Quantity of Tobacco Products Purchased in the Medium- and No-tax tiers - Product substitution (intensity and slope) | 1 day
  Purchasing of medium- and no-tax products in the ETM conditions will be fit to ordinary least squares regression for each tax tier. This yields slope measures of each tax tier's product purchasing, wherein more positive slopes indicate greater substitution (i.e., greater increases in purchasing of substitutes as tax magnitudes increase). Ordinary least squares regression is used here to model purchasing in the medium- and no-tax tier because it is capable of measuring positive slopes, indicative of substitution, and distinguishing these tiers from those that do not show substitution. In the event this relationship is non-linear, we will consider other relevant models.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Stein, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC; Christine E Sheffer, Ph.D., Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Fralin Biomedical Research Institute, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.